CLINICAL TRIAL: NCT04476784
Title: Clinical Assessment of a Daily Wear Monthly Replacement Soft Silicone Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLY935-C013
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-09

CONDITIONS: Myopia
Keywords: Contact lenses
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- LID018869, then Biofinity (Other): Lehfilcon A contact lenses worn first, followed by comfilcon A contact lenses, as randomized. Each product will be worn in both eyes during waking hours only for at least 5 days per week over a 30-day period. CLEAR CARE will be used for nightly cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Comfilcon A contact lenses; Device: CLEAR CARE
- Biofinity, then LID018869 (Other): Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each product will be worn in both eyes during waking hours only for at least 5 days per week over a 30-day period. CLEAR CARE will be used for nightly cleaning and disinfection.
  Interventions: Device: Lehfilcon A contact lenses; Device: Comfilcon A contact lenses; Device: CLEAR CARE

INTERVENTIONS:
Device: Lehfilcon A contact lenses — Investigational silicone hydrogel contact lenses
  Other Names: LID018869
Device: Comfilcon A contact lenses — Commercially available silicone hydrogel contact lenses
  Other Names: CooperVision® BIOFINITY®; Biofinity
Device: CLEAR CARE — Hydrogen peroxide-based cleaning and disinfecting solution

SUMMARY:
The purpose of this study is to assess the clinical performance of an investigational contact lens over 30 days of daily wear.

DETAILED DESCRIPTION:
Subjects will wear two products and be expected to attend 4 office visits. The individual duration of participation will be approximately 60 days (30 days for each product).

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an approved Informed Consent form;
* Willing and able to attend all scheduled study visits as required by the protocol;
* Current wearer of spherical weekly/monthly soft contact lenses in both eyes with at least 3 months wearing time of 5 days per week and 10 hours per day;
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Current or prior Biofinity contact lens wearer in the past 3 months;
* Monovision contact lens wearer;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2020-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research, LLC
Locations (5):
- United States (5):
  - Alcon Investigative Site, Maitland, Florida
  - Alcon Investigative Site, Bloomington, Illinois
  - Alcon Investigative Site, Pittsburg, Kansas
  - Alcon Investigative Site, Shawnee Mission, Kansas
  - Alcon Investigative Site, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 5 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all subjects/eyes (66/132) exposed to any study lenses evaluated in this study as treated (Safety Analysis Set)
Units Other Than Participants: eyes
Groups:
- LID018869, Then Biofinity: Lehfilcon A contact lenses worn first, followed by comfilcon A contact lenses, as randomized. Each product was worn in both eyes during waking hours only for at least 5 days per week over a 30-day period. CLEAR CARE was used for nightly cleaning and disinfection.
- Biofinity, Then LID018869: Comfilcon A contact lenses worn first, followed by lehfilcon A contact lenses, as randomized. Each product was worn in both eyes during waking hours only for at least 5 days per week over a 30-day period. CLEAR CARE was used for nightly cleaning and disinfection.
Period: First Wear Period (30 Days ± 2 Days)
Arm/Group | LID018869, Then Biofinity | Biofinity, Then LID018869
Started | 31; 62 eyes | 35; 70 eyes
Completed | 30; 60 eyes | 35; 70 eyes
Not Completed | 1; 2 eyes | 0; 0 eyes
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Wear Period (30 Days ± 2 Days)
Arm/Group | LID018869, Then Biofinity | Biofinity, Then LID018869
Started | 30; 60 eyes | 35; 70 eyes
Completed | 30; 60 eyes | 35; 70 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | LID018869, Then Biofinity | Biofinity, Then LID018869 | Total
Number analyzed (Participants) | 31 | 35 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (8.0) | 33.7 (8.7) | 33.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 35 | 66
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 30 | 34 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 35 | 66

OUTCOME MEASURES:

1. Primary Outcome: Mean Distance Visual Acuity (logMAR) With Study Lenses
Description: Visual acuity (VA) was collected for each eye individually with study lenses in place at a distance of 4 meters using a letter chart. VA was measured in logarithm minimum angle of resolution (logMAR). On Day 30, VA was assessed after 6-8 hours of wear. A logMAR value of 0 equates to 20/20 Snellen visual acuity (normal distance eyesight), with a lower logMAR value indicating better visual acuity. No formal hypothesis testing was planned.
Time Frame: Day 1, Day 30 after 6-8 hours of wear, each product
Population: Full Analysis Set: All randomized subjects who are exposed to any study lenses evaluated in this study.
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: eyes
Groups:
- LID018869: Lehfilcon A contact lenses worn in both eyes during waking hours only for at least 5 days per week over a 30-day period. CLEAR CARE was used for nightly cleaning and disinfection.
- Biofinity: Comfilcon A contact lenses worn in both eyes during waking hours only for at least 5 days per week over a 30-day period. CLEAR CARE was used for nightly cleaning and disinfection.
Arm/Group | LID018869 | Biofinity
Number analyzed (Participants) | 66 | 65
Number analyzed (eyes) | 132 | 130
logMAR
  Day 1 | -0.11 (0.08) | -0.13 (0.08)
  Day 30, after 6-8 hours of wear | -0.12 (0.07) | -0.13 (0.08)

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 60 days.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. The safety analysis set includes all subjects/eyes exposed to any study lenses evaluated in this study. For treatment-emergent safety analyses, subjects/eyes were categorized under the actual study lenses exposed in the corresponding lens sequence.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID018869 - Ocular; LID018869 - Nonocular: Events reported in this group occurred while exposed to lehfilcon A contact lenses
- Biofinity - Ocular; Biofinity - Nonocular: Events reported in this group occurred while exposed to comfilcon A contact lenses
Arm/Group | Pretreatment | LID018869 - Ocular | LID018869 - Nonocular | Biofinity - Ocular | Biofinity - Nonocular
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/130 | 0/65
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/130 | 0/65
Other Adverse Events (participants affected / at risk) | 0/66 | 0/132 | 0/66 | 0/130 | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-07-09): https://cdn.clinicaltrials.gov/large-docs/84/NCT04476784/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT04476784/SAP_001.pdf